CLINICAL TRIAL: NCT00614315
Title: A Prospective Observational Study of the FLAIR™ Endovascular Stent Graft Optimized Delivery System
Brief Title: FLAIR™ Delivery System Study
Acronym: FLAIR DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-07-001
Record Dates: First submitted 2007-12-18; First posted 2008-02-13 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Constriction, Pathologic
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLAIR Endovascular Stent Graft and Delivery System (Experimental)
  Interventions: Device: FLAIR™ Endovascular Stent Graft

INTERVENTIONS:
Device: FLAIR™ Endovascular Stent Graft — The FLAIR™ Endovascular Stent Graft is designed to treat venous anastomotic stenoses of AV access grafts, providing both structural support of the site following angioplasty (stent), and a barrier to locally recurrent flow-limiting neointimal tissue growth (covering/graft).

SUMMARY:
The objective of this clinical study is to evaluate the performance of the Optimized FLAIR™ Delivery System.

ELIGIBILITY:
Inclusion Criteria:

* The subject is either a male or non-pregnant female ≥ 18 years old.
* The subject has been properly informed about the study per IRB requirements, and has signed and dated the IRB-approved ICF.
* The subject is willing to comply with the protocol requirements and can be contacted by telephone.
* The subject has a synthetic AV access graft located in an arm that has been implanted for > 30 days and has undergone at least one successful dialysis session prior to the index procedure.
* Angiographic evidence indicates that the subject has a stenosis of >50% located at the graft-vein anastomosis of the subject's synthetic AV access graft.
* The target lesion is estimated to be ≤ 7 cm in length by angiography prior to performance of any interventional procedures.
* The entire target lesion is located within 7 cm of the graft-vein anastomosis, as verified by angiography, such that approximately 1 cm of the FLAIR™ Endovascular Stent Graft will extend into non-diseased vein and approximately 1 cm but no more than 2 cm of the FLAIR™ Endovascular Stent Graft will extend into non-diseased AV graft.
* Graft diameter at the deployment site is between 5 mm and 8 mm, as verified by angiography.
* Full expansion of an appropriately sized angioplasty balloon, in the operator's judgment, can be achieved during primary angioplasty.

Exclusion Criteria:

* The subject has a life expectancy of < 6 months.
* The presence of a previously placed stent and/or stent graft located in the treatment area. The treatment area is defined as the entire target lesion and 1 cm of landing zone into both non-diseased AV graft and non-diseased vein.
* The subject has an infected AV access graft or other infection.
* The location of the target lesion would require that the FLAIR™ Endovascular Stent Graft be deployed fully across the elbow joint.
* The location of the target lesion would require that the FLAIR™ Endovascular Stent Graft cross an angle (between the outflow vein and synthetic AV access graft) that is > 90 degrees.
* The subject has an uncorrected blood coagulation disorder.
* The subject has a known allergy or sensitivity to contrast media which cannot be adequately pre-medicated.
* Subject is currently enrolled or scheduled to be enrolled in other investigations that conflict with follow-up testing or confounds data in this trial.
* The subject has a known hypersensitivity to nickel-titanium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Rosenblatt, M.D., Principal Investigator — Connecticut Image Guided Surgery
Locations (1):
- Connecticut Image Guided Surgery, Fairfield, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FLAIR Endovascular Stent Graft: Patients treated with the FLAIR Endovascular Stent Graft
Period: Overall Study
Arm/Group | FLAIR Endovascular Stent Graft
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FLAIR Endovascular Stent Graft
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (15.14)
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Technical Success for Delivery
Description: defined as deployment of the implant to the intended location, assessed at the time of the index procedure.
Time Frame: Measured at the time of implantation (Day 0)
Measure: Number; unit: Percentage of successful implantations
Arm/Group | FLAIR Endovascular Stent Graft
Number analyzed (Participants) | 30
Percentage of successful implantations | 100

2. Secondary Outcome: Number of Device/Procedure-related Adverse Events(Safety of Delivery)
Description: Device/Procedure-related adverse events from the index procedure through 30 days post procedure
Time Frame: Index Procedure to 30 days
Measure: Number; unit: Number of Device/Procedure events
Arm/Group | FLAIR Endovascular Stent Graft
Number analyzed (Participants) | 30
Number of Device/Procedure events | 1

ADVERSE EVENTS:
Time Frame: 30 days post implantation
Arm/Group | FLAIR Endovascular Stent Graft
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLAIR Endovascular Stent Graft (N=30)
Thrombosis of Access Circuit (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No